CLINICAL TRIAL: NCT01860105
Title: Appraisal of MDCO-157 and Plavix® Pharmacokinetics and Pharmacodynamics in Healthy Volunteers With an Open-label, Randomized, Cross-over Evaluation: The AMPHORE Study
Brief Title: Appraisal of MDCO-157 and Plavix® Pharmacokinetics and Pharmacodynamics in Healthy Volunteers With an Evaluation
Acronym: AMPHORE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-157-12-01
Record Dates: First submitted 2012-09-12; First posted 2013-05-22 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pharmacokinetics and Pharmacodynamics in Healthy Volunteers
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 75mg MDCO-157 (Active Comparator): iv
  Interventions: Drug: MDCO-157
- 150mg MDCO-157 (Active Comparator): iv
  Interventions: Drug: MDCO-157
- 300mg MDCO-157 (Active Comparator): iv
  Interventions: Drug: MDCO-157
- 300mg PLAVIX (Active Comparator): oral
  Interventions: Drug: PLAVIX

INTERVENTIONS:
Drug: MDCO-157 — intravenous administration
  Arms: 150mg MDCO-157; 300mg MDCO-157; 75mg MDCO-157
Drug: PLAVIX — oral administration
  Arms: 300mg PLAVIX

SUMMARY:
Following a first, dose ascending study that enrolled 144 normal healthy volunteers (NHVs), this study, to be conducted in approximately 36 NHVs, will provide pertinent information in determining the dose-response of MDCO-157 for platelet aggregation inhibition and P2Y12 receptor inhibition effects and in selection of doses that match the antiplatelet effects of 300 mg PLAVIX® ®. The study will also provide additional data for pharmacokinetics (PK), safety and tolerability of single doses of MDCO-157.

ELIGIBILITY:
Inclusion Criteria

* Healthy males or females 18 to 45 years of age, inclusive.
* Provide written informed consent for genetic testing and written informed consent for the study before initiation of any study related procedures
* Affiliated to the French social security system
* Screening and baseline Fridericia's correction (QTcF) interval < 450 msec and baseline heart rate between 50 and 100 bpm (inclusive)

Exclusion Criteria:

* Known or suspected hypersensitivity or allergy to clopidogrel, Captisol, PLAVIX® , or its excipients
* Body mass index <20 or > 30 kg/m²
* Inability to communicate with the investigator or comply with study related procedures, or high likelihood of being lost to follow up
* Known or suspected pregnancy or lactating female
* Medical history, physical examination including 12-lead ECG or laboratory evaluation conducted at the screening visit with results indicative of any disease or condition which might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Tobacco product use within the last 6 months prior to dosing
* Platelet count < 150,000/µL
* A personal or family history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations
* Active pathological bleeding such as peptic ulcer or intracranial hemorrhage
* Positive screen for Hepatitis B (Hepatitis B Surface Antigen HBsAg), Hepatitis C (Hepatitis C Antibody), or HIV (anti-HIV 1/2)
* Received an investigational drug within a period of 30 days or 5 half-lives, whichever is longer, prior to enrollment in the study
* Use of aspirin, other non-steroidal anti-inflammatory drugs, CYP3A4 inhibitors (ketoconazole), CYP2C19 inhibitors (eg, omeprazole) or other drugs known to affect platelet function or coagulation within 14 days prior to receiving study drug (MDCO-157 or oral clopidogrel)
* Grapefruit within 10 days prior to receiving study drug (MDCO-157 or PLAVIX®)
* Use of any over-the-counter medication, including herbal products, within 7 days prior to administration of study drug (MDCO-157 or PLAVIX®), except for up to 2 grams of acetaminophen per day for up to 3 days for pain control

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Dose Response of MDCO-157 (3 doses) compared to Plavix 300 mg | 24 hr
  To evaluate the dose-response of MDCO-157 (at 3 doses) compared to Plavix (300 mg), using Emax and AUEC with VASP, over 24 hours:
  * Maximum effect of P2Y12 receptor inhibition (Emax) using VASP (flow cytometry)
  * Area under the effect of P2Y12 receptor inhibition time curve (AUEC) using VASP (flow cytometry)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of MDCO-157 and its metabolites | 24 hrs
  To determine the pharmacokinetic (PK) of MDCO-157, including clopidogrel, clopidogrel carboxylic acid, and clopidogrel H4 thiol active metabolite in plasma
Safety and tolerability | 48 hrs post each treatment period
  To assess the safety and tolerability of single doses of MDCO 157 (75 mg, 150mg and 300mg) as measured by assessment of AEs and SAEs.
Dose response of MDCO-157 as assessed by LTA | 24 hours
Dose response of MDCO-157 as assess by VerifyNow P2Y12 assay | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Collet JP, Funck-Brentano C, Prats J, Salem JE, Hulot JS, Guilloux E, Hu MY, He K, Silvain J, Gallois V, Brugier D, Anzaha G, Galier S, Nicolas N, Montalescot G. Intravenous Clopidogrel (MDCO-157) Compared with Oral Clopidogrel: The Randomized Cross-Over AMPHORE Study. Am J Cardiovasc Drugs. 2016 Feb;16(1):43-53. doi: 10.1007/s40256-015-0145-0. PMID 26386578